CLINICAL TRIAL: NCT06803420
Title: AI-powered Portable MRI Abnormality Detection
Acronym: APPMAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRAS 347453
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Head Injury
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Portable, ultra-low-field MRI scanner (Experimental): Patients undergoing a standard brain MRI scan will be invited to have an additional portable MRI scan within 30 days of their clinical scan.
  Interventions: Device: Portable, ultra-low-field MRI scanner

INTERVENTIONS:
Device: Portable, ultra-low-field MRI scanner — This study evaluates a portable, ultra-low-field MRI scanner (the Hyperfine Swoop) combined with artificial intelligence (AI) to detect brain abnormalities.
  Patients undergoing a standard brain MRI scan will be invited to have an additional portable MRI scan within 30 days of their clinical scan. The portable MRI scan will take approximately 60 minutes, using multiple imaging sequences, including T2-weighted scans.
  The AI system will then analyse the portable MRI images and categorise them as "normal" or "abnormal". The results will be compared with expert neuroradiologist reports from standard MRI scans to validate accuracy.
  This intervention aims to assess whether portable MRI with AI can provide a low-cost, accessible alternative to standard MRI, potentially improving triage and reducing waiting times for patients requiring urgent brain imaging.

SUMMARY:
This study aims to test a new AI-powered portable MRI scanner that can quickly identify whether a brain scan is normal or abnormal. Currently, standard MRI scans are expensive and have long waiting times. Our goal is to see if a smaller, cheaper, and more accessible MRI scanner-combined with artificial intelligence (AI)-can help doctors identify abnormalities faster and improve patient care.

We will invite patients from King's College Hospital (KCH) who are already having a standard MRI scan. They will be asked to have an extra scan using the portable MRI, which takes about 60 minutes. The AI tool will then analyse these scans and compare its results to those of expert radiologists.

By the end of the study, we hope to prove whether portable MRI with AI can be used in hospitals and GP clinics, making brain scans more accessible, reducing wait times, and helping doctors prioritise urgent cases.

This study is funded by the Medical Research Council (MRC) and has been approved by UK research ethics committees.

ELIGIBILITY:
Inclusion Criteria:

Adults ≥18 years old. Undergoing standard brain MRI including T2-weighted sequences.

Exclusion Criteria:

Contraindications to MRI (e.g. pacemaker, pregnancy). Poor quality MRI scans without a neuroradiology report.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Accuracy of AI toll for triaging scans as "normal or "abnormal" | 36 months
  Ai Triage accuracy compared with consultant neuroradiologists assessment.

SECONDARY OUTCOMES:
Generalisability of AI tool (evaluated on external dataset). | 36 months
Patient acceptability of portable MRI (survey/interviews) | 36 months
Feasibility of integrating portable MRI in clinical pathways. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Booth, Dr, Principal Investigator — King's College London & King's College Hospital

IPD SHARING:
Plan to Share IPD: No